CLINICAL TRIAL: NCT05275283
Title: Efficacy Evaluation of Positive End-expiratory Pressure in Children Undergoing Mechanical Ventilation Using Supraglottic Airway Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2111-073-1272
Record Dates: First submitted 2021-11-29; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Positive End Expiratory Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Applying tidal volume 7 ml/kg without PEEP
- PEEP group (Experimental): Applying tidal volume 7 ml/kg with 6 cmH2O of PEEP
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — 6 cmH2O of PEEP
  Arms: PEEP group

SUMMARY:
The aim of this study is to determine whether application of positive end-expiratory pressure (PEEP) improves respiratory data including respiratory compliance in children who receive positive pressure ventilation using supraglottic airway device (SAD).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 6 years of age who are scheduled simple operation under general anesthesia
* SAD was used for mechanical ventilation

Exclusion Criteria:

* Abdominal distension, risk of pulmonary aspiration
* Bronchopulmonary dysplasia/respiratory distress syndrome
* Pneumothorax
* Airway surgery
* Thoracic surgery or laparotomy
* Surgery under prone position

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory system compliance | at the end of surgery, about 2 hours after starting of mechanical ventilation
  total lung and chest wall compliance, ml/cmH2O

SECONDARY OUTCOMES:
Respiratory system compliance | 10 minutes, 30 minutes, 60 minutes after starting of mechanical ventilation
  total lung and chest wall compliance, ml/cmH2O
oropharyngeal leak pressure | immediate after SAD insertion
  cmH2O
Electrical impedance tomography parameter - dynamic compliance | throughout anesthesia (about during 1-3 hours)
  ventilation/airway pressure (cmH2O)
Electrical impedance tomography parameter - regional ventilation delay | throughout anesthesia (about during 1-3 hours)
  assessment of ventilation homogeneity (no unit)
Electrical impedance tomography parameter - pulmonary opening pressure | throughout anesthesia (about during 1-3 hours)
  pressure requiring opening of alveoli (cmH2O

CONTACTS AND LOCATIONS:
Locations (1):
- Hee-Soo Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided